CLINICAL TRIAL: NCT02661724
Title: Take Charge of Burn Pain: A Randomized Controlled Trial of a Web-based Self-Management Intervention to Improve Burn Pain Outcomes
Brief Title: Take Charge of Burn Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The Phoenix Society for Burn Suvivors (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00054201
Record Dates: First submitted 2016-01-13; First posted 2016-01-22 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Burn Related Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Take Charge Burn - Pain (TCBR-Pain) (Experimental): The TCBR-Pain program includes 7 lessons addressing key dimensions of pain management for persons with burn injury. Each session is about 20 minutes and focuses on burn injury recovery and life style education. Sessions begin with a brief self-assessment and in later sessions, the participant is given graphical feedback on their progress.
  Interventions: Behavioral: TCBR-Pain
- Education attention control (No Intervention): The attention group receives an educational materials that is matched to the TCBR-Pain intervention in terms of session length and time on the web-based program. The web-based Education attention condition includes 7 sessions delivered over 7 weeks. The Education Attention Control is education materials commonly employed in rehabilitation centers and has been successfully used in several studies as a comparison to active rehabilitation interventions

INTERVENTIONS:
Behavioral: TCBR-Pain — The interactive TCBR-Pain uses programmed learning, skill development and behavioral practice to engage persons with burn pain in self-management of pain and related problems. The TCB-Pain program includes 7 lessons addressing key dimensions of pain management for persons with burn injury. Each session is about 20 minutes and focuses on burn injury recovery and life style education. Sessions begin with a brief self-assessment and in later sessions, the participant is given graphical feedback on their progress. The lessons are narrated and include closed captioning, are animated, and include branching to provide personalized content.
  Arms: Take Charge Burn - Pain (TCBR-Pain)

SUMMARY:
Persons with burn-related pain remain under treated and do not have access to comprehensive burn pain management. We seek to extend evidence-based cognitive behavioral pain management strategies to a group of burn survivors that are currently under treated for for burn pain with a specific goal of reducing pain related interference in life activities.

Investigators will conduct a randomized controlled trial to test the central hypothesis that a computer-based cognitive-behavioral program (Take Charge of Burn Pain) will improve pain management, psychological health, and improve participation in burn survivors. Specific aims include: 1) to determine the efficacy of a web-based self-management intervention in reducing pain and pain-related interference and increasing pain management self-efficacy; and 2) to determine whether Take Charge of Burn Pain improves psychological health and participation in life activities in persons with burn injury pain. Emerging research suggests that web-based pain management interventions may be a feasible and effective alternative to clinic-based interventions for patients with mobility and geographic restrictions, such as those treated at tertiary burn centers.

DETAILED DESCRIPTION:
Burns are among the most painful of all injuries requiring painful daily wound care and rehabilitation procedures. Despite the best efforts of burn care professionals, burns frequently result in acute and chronic suffering and poor functional outcomes for otherwise healthy individuals with many years of productive life remaining. The evidence base directing burn pain management is generally weak, with much work based on clinical preferences rather than scientific evidence. There is a tremendous need for clinical trials to evaluate and improve the standard of care. While pharmacological treatment options are widely available for burn survivors throughout the emergent, acute, and rehabilitation phases of healing there is limited access to comprehensive pain management. It is critical to establish accessible pain management approaches that address the emotional, cognitive and physical dimensions of the burn pain experience. Cognitive behavioral therapy (CBT) has proven effective for patients with chronic pain and studies have demonstrated the efficacy of providing tele-rehabilitation CBT services for improving outcomes in persons with disability. However, tele-rehabilitation CBT pain management has not been traditionally offered or studied in persons with burn-related pain. The population of burn survivors has limited access to comprehensive pain management including CBT due to lack of access, financial constraints, and mobility issues that render clinic-based CBT impractical. Innovative rehabilitation interventions and delivery methods are needed to improve pain, functional, psychological and participation outcomes in burn survivors with significant, yet untreated, pain problems.

Investigators propose to conduct a two group randomized controlled trial to test the central hypothesis that web-based CBT will improve pain severity, pain interference, self-efficacy, psychological health and participation in life activities for burn survivors with pain. Emerging research suggests that tele-rehabilitation may be a feasible, and effective alternative (with much broader applicability) to clinic-based interventions for patients with access restrictions. This project will address 2 specific aims:

Specific Aim 1: To determine the efficacy of a web-based, CBT self-management intervention (Take Charge of Burn Recovery - Pain [TCBR-Pain) in improving pain management self-efficacy, and reducing pain and pain-related interference in burn survivors with pain.

Outcomes will be measured using a battery of standardized tests at baseline, 2 month (treatment completion) and 5 month post-treatment follow-up. Self-reported pain self-efficacy, pain severity and pain interference will be measured using validated instruments (Pain Self-efficacy Scale, Brief Pain Inventory respectively).

Hypothesis 1: TCBR- Pain participants will demonstrate significantly greater improvement in pain self-efficacy, pain severity and pain interference relative to the attention-control group at 2 month (treatment completion) and 5 month follow up.

Specific Aim 2: To determine the efficacy of a web-based, CBT self-management intervention ((Take Charge of Burn Recovery - Pain [TCBR - Pain]) for improving psychological health and participation in life activities for burn survivors with pain.

Outcomes will be measured using a battery of standardized tests at baseline, 2 month (treatment completion) and 5 month follow-up. Self-reported depression and anxiety, and participation in life activities will be measured using validated instruments (PHQ-9 Depression Scale and PCL -Civilian Anxiety Scale, and the World Health Organization Disability Assessment Scales [WHODAS-II]) respectively.

Hypothesis 2: TCBR- Pain participants will demonstrate significantly greater improvement in depressive and anxiety symptoms and participation relative to the attention-control group at 2 month (treatment completion) and 5 month follow up.

This initial randomized trial will provide critical data on recruitment and retention as well as effect sizes and sample sizes for in the next stage of research - a multi-center, clinical trial which will determine scalability of the intervention. In the proposed study, we will consent 256 burn survivors with pain and randomly assign them to the intervention or control group. After informed oral consent is obtained, potential participants will be screened for eligibility. If eligible, (see inclusion/exclusion criteria below) participants will be consented and will complete the baseline assessment on-line. Once the web-based assessment is complete, the participants will be randomly assigned to either the web-based 7 lesson TCBR - Pain program or the 7 lesson Attention Control -Education group. Randomization will occur in balanced blocks to stratify group composition by pain level, self-reported Total Burn Surface Area, and time since initial burn injury. Participants will complete the post-intervention assessment at 2 months and again at 5 months to assess pain severity, pain interference, psychological health, and participation in life activities. Participants who obtain other treatments while enrolled in the study will be included and these other interventions will be documented and controlled in analyses if necessary. Findings from this study will support future research and dissemination efforts to improve the pain management, psychological health and life participation of patients following burn injury through innovative rehabilitation interventions and delivery methods.

ELIGIBILITY:
Inclusion Criteria:

1. Persons ages 18 to 70 years old having experienced a burn injury requiring hospitalization at least 6 months prior to enrollment;
2. Reporting a pain severity score on the Brief Pain inventory of 4 (0-10) or higher;
3. Reporting pain of at least 3 months duration; and
4. English speaking due to feasibility of providing the web-based intervention only in English at this time.

Exclusion Criteria:

1. Significant neurological or psychiatric condition precluding informed consent.
2. Lack of access to a computer that is connected to the worldwide web.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2015-04; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain Severity and Pain-Related Interference | 2 and 5 month
  The Brief Pain Inventory (BPI) will be used to assess pain severity and establish that the pain intensity inclusion criteria are met. The BPI includes two primary dimensions: pain severity (4 items) and pain interference (7 items), each rated on 0 to 10 scales.

SECONDARY OUTCOMES:
Change in Depression | 2 and 5 month
  Depression and PTSD Anxiety will be measured using the Patient Health Questionnaire-9 (PHQ-9) . In a psychometric study of the PHQ-9, the instrument demonstrated acceptable test-retest reliability and was both sensitive (0.93) and specific (0.89) when compared to a diagnosis of major depression in persons with traumatic injury.
Change in Participation in life activities | 2 and 5 month
  Participation in life activities will be measured using the World Health Organization Disability Assessment Scales (WHODAS-II) is a 36-item general disability instrument that has been specifically designed to use the ICIDH-2 framework to evaluate the dimensions of disability- activity and participation.
Change in PTSD Anxiety | 2 and 5 month
  PTSD Checklist-Civilian Version (PCL-C). The PCL-C has demonstrated acceptable test-retest reliability and internal consistency values and good convergent validity with moderate to high correlations with other PTSD instruments and measures of anxiety and depression in persons with traumatic injury. Studies have also found that trauma survivors with PCL-C scores ≥ 45 have a greater than 75% probability of developing symptoms consistent with a diagnosis of PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wegener, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staguhn ED, Kirkhart T, Allen L, Campbell CM, Wegener ST, Castillo RC. Predictors of participation in online self-management programs: A longitudinal observational study. Rehabil Psychol. 2024 May;69(2):102-109. doi: 10.1037/rep0000521. Epub 2023 Nov 13. PMID 37956087